CLINICAL TRIAL: NCT07263178
Title: A Multi-center, Prospective, Observational Study to Assess the Treatment Patterns and Prognosis of Second and Later-line Palliative Chemotherapy in Patients With Metastatic Colorectal Cancer Who Failed First-line Palliative Chemotherapy
Brief Title: A Study of Second- and Later-line Palliative Chemotherapy in Patients With Metastatic Colorectal Cancer.
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-CPT-OS-402
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Palliative chemotherapy; Metastatic Colorectal Cancer; Observation Study
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Second and later-line palliative chemotherapy — As this is a non-interventional study designed to collect data as part of routine clinical practice, the selection and dosage of medication, treatment period, and whether or not to change it are all based on the clinician's judgment

SUMMARY:
This study aims to comprehensively identify the various treatment patterns of second- or subsequent-line palliative chemotherapy used in patients with metastatic colorectal cancer who have experienced failure of first-line palliative chemotherapy and to evaluate the prognosis of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent after receiving information about the purpose and method of this study.
* Patients with histologically and radiologically confirmed metastatic colorectal cancer (colorectal cancer) who have evaluable (measurable) lesions.
* Patients scheduled to receive their first second-line palliative chemotherapy following failure of first-line palliative chemotherapy (including those who relapse during or within 6 months after completion of postoperative adjuvant therapy, necessitating palliative chemotherapy).
* Patients who understand the research, are cooperative in the research process, and are deemed capable of participating until the completion date.

Exclusion Criteria:

* Female patients who are pregnant, have childbearing potential, or are breastfeeding.
* Has received an investigational product within 4 weeks from the study enrollment or has plans to participate in another clinical trial during the participation of this study.
* Other subjects who are considered inappropriate to participate in this study by the judgment of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer (colon and rectal cancer) who have failed first-line palliative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Progression-free survival (PFS) by treatment pattern

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months
  Overall Survival (OS) by treatment pattern
Dosage period for each treatment pattern | up to 24 months
Objective Response Rate (ORR) | up to 24 months
Types of Secondary palliative chemotherapy | up to 24 months
Types of Third palliative chemotherapy | up to 24 months
Conversion rate | up to 24 months
  Conversion rate to resectable group by treatment pattern
Quality of Life Assessment | up to 12 months
  The FACT-C (Functional Assessment of Cancer Therapy-Colorectal) questionnaire uses a 5-point Likert-type scale. The responses generally range from 0 (Not at all) to 4 (Very much).
Eastern Cooperative Oncology Group Performance Status(ECOG PS) Assessment | up to 24 months
  The ECOG PS uses a scale from 0 to 5, where a score of 5 specifically means the patient is deceased. The score of 0 indicates the best performance status (fully active), while 4 indicates the worst performance status for a living patient (completely disabled/bedridden).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea